CLINICAL TRIAL: NCT05456139
Title: Effectiveness Trial of the Early Social Interaction (ESI) Model Using Mobile Technology for Toddlers With Autism Identified From Early Screening in Primary Care
Brief Title: Effectiveness Trial of Mobile ESI for Toddlers With Autism Identified by Early Screening in Primary Care
Acronym: ESI-MC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy M. Wetherby, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00002656; R01MH121627 (NIH); R01MH121622 (NIH); R01MH127120 (NIH)
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Pediatrics; Telehealth; Treatment; Early Intervention; Community-based
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The investigators will conduct an effectiveness trial of ESI-MC to address the question of whether starting evidence-based intervention earlier leads to better outcomes than starting later. The investigators will address this question by using a modified stepped wedge design and blended implementation research to analyze data obtained with ESI-MC start at 18, 24, or 30 months. he investigators will diagnostically ascertain 240 children from a pool of 360 18-month-olds with early signs of autism. The 240 children will be randomly assigned to one of three ESI-MC timing groups. The investigators will measure child active engagement and social communication change every 6 months as the primary outcome variables. Outcome measures of developmental level, autism symptoms, and adaptive behavior will be examined to measure differential treatment effects.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigator and diagnosticians will be kept blind to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual Only (Active Comparator): During 2 of the 3 six-month periods of participation, families will receive Treatment as Usual (TAU) only. Families in the TAU control condition will receive usual care and EI service in their community, which will be tracked with the BSRC Intervention History Form. Because all families join My Baby Navigator and will be screened by the SoCo CheckUp, families in both conditions will have access to the "Seamless Path for Families" which includes online tools about social communication developmental milestones. Families will also have access to Autism Navigator About Autism in Toddlers, the ASD Video Glossary, and the Autism Navigator How-to Guide for Families, a self-guided online course.
  Interventions: Behavioral: Treatment as Usual
- ESI-MC plus Treatment as Usual (Active Comparator): During 1 of the 3 six-month periods of participation, families will receive 24 weekly sessions of Early Social Interaction via Mobile Coaching (ESI-MC) by a trained early intervention provider. ESI-MC is an evidence-based parent-implemented intervention for toddlers with ASD. ESI teaches parents how to support their child's social communication, language, play and behaviors in everyday routines, activities, and places. Program planning entails building consensus with families on priority targets for the child and teaching strategies and supports for the parents using manualized conversational steps, Baby Navigator social communication milestones, and ESI content for families to practice 25 hours per week. Families will be invited to participate in the online Autism Navigator How-To Guide, a self-guided web-based course and companion online group education meetings. Families will also receive Treatment as Usual (TAU).
  Interventions: Behavioral: Early Social Interaction Mobile Coaching (ESI-MC)

INTERVENTIONS:
Behavioral: Treatment as Usual — Families in the Treatment as Usual (TAU) condition will receive usual care and EI services in their community, which will be tracked with the BSRC Intervention History Form. Because all families join My Baby Navigator and will be screened by the SoCo CheckUp, families in both conditions will have access to the "Seamless Path for Families" which includes online tools about social communication developmental milestones. Families will also have access to Autism Navigator About Autism in Toddlers, the ASD Video Glossary, and the Autism Navigator How-to Guide for Families, a self-guided online course.
  Arms: Treatment as Usual Only
Behavioral: Early Social Interaction Mobile Coaching (ESI-MC) — The ESI-MC coach will offer 24 weekly sessions for the 6-month ESI-MC condition. The parent will be the focus of training. Each session includes: setting the stage to develop that session's agenda; intervention implementation with these coaching steps: a) review the target, b) use guided/caregiver practice, or video review to teach the strategy, c) provide specific feedback to support caregiver reflection and independence in the activity, and d) problem solving and plan for next time; steps a-d are repeated for 3-5 activities per session; and summarize plans for deliberate practice between sessions. Families will be invited to participate in the online Autism Navigator How-To Guide, a self-guided online course and companion to the online group education meetings to engage families in the content of the online course and provide support through interaction with other families. Families will also participate in TAU usual care and EI services in their community.
  Arms: ESI-MC plus Treatment as Usual

SUMMARY:
The goal of this collaborative R01 is to demonstrate the therapeutic value and community-wide implementability of an early intervention (EI) platform for toddlers with autism spectrum disorder (ASD) that is completely virtual, from recruitment through intervention. This platform-Early Social Interaction Mobile Coaching (ESI-MC) deploys individual telehealth sessions with coaching and feedback to help families embed intervention in everyday activities. Specifically, the investigators will conduct an effectiveness trial of ESI-MC to address the important question of whether starting evidence-based intervention earlier leads to better outcomes than starting later. The investigators will address this question by using a modified stepped wedge design and blended implementation research to analyze data obtained with ESI-MC start at 18, 24, or 30 months. The investigators will diagnostically ascertain 240 children from a pool of 360 18-month-olds with early signs of autism, 30 in each of 8 US regions (Central and SW Florida; Atlanta, GA; suburbs of Philadelphia, PA; New York City, NY; Cincinnati, OH; Chicago, IL; Seattle, WA; and Los Angeles, CA). Research participants will be recruited using a new virtual platform-My Baby Navigator-linking a new surveillance and screening tool, an app to upload video-recorded home observations and telehealth intervention sessions, and a package of educational resources. The 240 children will be randomly assigned to one of three ESI-MC timing groups. ESI-MC will be delivered by community-based early intervention providers (EIPs) currently working within the the early intervention system in the recruitment regions. The investigators will measure child active engagement and social communication change every 6 months as the primary outcome variables. Outcome measures of developmental level, autism symptoms, and adaptive behavior will be examined to measure differential treatment effects. Maximizing the use of mobile technology, ESI-MC offers the prospect of a community-viable, scalable and sustainable treatment to improve EI services for toddlers with ASD, particularly among minority and low-resource communities.

DETAILED DESCRIPTION:
This is a collaborative R01 application (RFA-MH-18-700) with Dr. Amy Wetherby as PI at Florida State University (FSU), Drs. Ami Klin and Jennifer Stapel-Wax as Co-PIs at Emory University (EU), and Dr. Catherine Lord as Co-PI at the University of California, Los Angeles (UCLA). This effectiveness trial will address the important question of whether starting evidence-based intervention earlier leads to better outcomes than starting later. The investigators will compare the timing of Early Social Interaction Mobile Coaching (ESI-MC) -individual telehealth sessions with coaching and feedback to help families embed intervention in everyday activities, starting at 18, 24, or 30 months, with a modified stepped wedge design and blended implementation research. This effectiveness trial will be conducted using a virtual platform from recruitment through intervention implementation to reach a national community-based sample of toddlers with autism spectrum disorder (ASD).

Overview of Effectiveness Trial. The investigators will recruit 360 children with early signs of autism at 18 months using a new virtual platform-My Baby Navigator-linking surveillance and screening tools, an app for uploading video-recorded home observations and mobile intervention sessions, and a package of educational resources. From the pool of 360 children with early signs, the investigators will identify 240 children with a clinical best estimate diagnosis of ASD, 60 in each of four regions (Northeast, Southeast, Midwest, West Coast), and randomly assign parent-child dyads to one of three ESI-MC timing groups (18, 24, 30) to address the following research aims:

Aim 1. Compare the effectiveness of ESI-MC implemented for 6 months on proximal outcome measures of child active engagement, child social communication change, parent transactional supports, and parent evidence-based strategy use (1A) with Treatment-as-Usual (TAU) at 24 and 30 months and (1B) across treatment timing groups initiated at 18, 24, or 30 months. Hypotheses 1) Parent-child dyads in ESI-MC will (1A) show significantly better child and parent outcomes compared to TAU and (1B) those starting ESI-MC earlier will show successively better child outcomes than those starting later.

Aim 2. Examine (2A) change in parent transactional supports and evidence-based strategy use as the mechanism for change in proximal child outcomes and (2B) individual child and family characteristics that moderate response to treatment.

Aim 3. Compare the effectiveness of ESI-MC implemented for 6 months on secondary outcome measures of child developmental level, autism symptoms, and adaptive behavior (3A) with TAU at 24 and 30 months and (3B) across treatment timing groups initiated at 18, 24, or 30 months.

Aim 4. Explore outcomes at 36 months, individual patterns of change from 18-36 months, and predictors of change across treatment timing groups by estimating child growth trajectories.

Aim 5. Examine barriers and promotive factors impacting widespread dissemination, implementation and sustainability across racial, socioeconomic and geographic lines, including parental uptake, engagement and satisfaction during and after intervention, treatment fidelity, reduction of disparities in access to services and in outcomes, and cost-benefit analyses.

The investigators expect ESI-MC will result in better outcomes than TAU and that initiating treatment earlier leads to better outcomes. This effectiveness trial of ESI-MC will address concerns raised by the US Preventive Services Task Force (USPSTF), advance knowledge for community-uptake, and provide needed evidence to support early universal screening and referral at 18-24 months. Documenting the therapeutic value of ESI-MC to teach parents in natural environments will offer a community-viable and affordable treatment to improve services for toddlers with ASD, which in light of ongoing COVID-19 pandemic restrictions, places a premium on remote tools and methods. The recent spotlight on healthcare disparities and civil injustices underscores the urgency with which inequalities faced by minority and low-resource communities need to be vigorously addressed. By maximizing the use of mobile technology and community-based care teams, this treatment will be ready for immediate, rapid, scalable, and sustainable deployment across the US that can lead to transformative changes in healthcare services for toddlers with autism and their families.

Overview of Collaborative Study. A collaborative study is necessary to accommodate a large, representative community-based sample of very young children with ASD with geographic spread for an effectiveness trial. Recruitment and implementation across 8 sites in 4 national regions will provide racial/ethnic and socioeconomic diversity, ample urban/rural areas, and different health service systems. The research team includes the complementary expertise needed and has history of collaboration. The PIs will establish a means of coordinating communication and shared decision-making before the start of research. FSU will provide the virtual platform for recruitment and random assignment, train the ESI mobile coaches, monitor intervention fidelity, and oversee data management and statistical analysis. UCLA will oversee reliability of autism symptom measures and calibration of diagnosis. Emory will oversee documentation and dissemination of research-based solutions to address health disparities. Each site will conduct diagnostic evaluations, ensure reliability on measures, and use manualized procedures conducted with fidelity to ensure scientific integrity for pooling data.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) complete the SoCo CheckUp by the time the child is 18 months of age and results will indicate positive risk for autism
* Parent(s) submit a home observation video of the parent engaging their child for an hour in 6 everyday activities by the time the child is 18 months of age
* Results of the SORF rated from the home observation indicate risk for autism
* The child receives a clinical best estimate diagnosis of autism spectrum disorder based on a diagnostic and developmental evaluation by 18 months (+/-2 months) of age, which includes completion of the ADOS
* The child will have sufficient trunk stability and control of arm and hand movements to hold objects and make simple gestures (give, show, reach)
* Parent(s) agree to be in the intervention study by the time the child is 18 months (+/- 2 months) of age
* The primary language at home is English or Spanish (the SoCo CheckUp and all Baby Navigator tools are available in these languages)
* The family lives within 45 miles of one of the 8 recruitment sites.

Exclusion Criteria:

* Child does not meet diagnostic criteria for autism
* Family does not agree to be video recorded
* Family does not agree to receive the intervention via mobile technology
* Enrollment in EI at the time of screening
* A sibling is already enrolled in the trial
* Children with significant motor, visual, or hearing impairments
* Children born with very low birth weight or significant medical complications (e.g., seizure disorder)

Ages: 15 Months to 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Parent-Child Interaction Change at Home | Baseline and 3, 6, 9, 12, 15, and 18 months thereafter
  Parent use of responsive learning strategies and child active engagement will be periodically assessed using the Measure of Active Engagement and Transactional Supports (MAETS). The MAETS is a rating of a video-recorded home observation of parent-child interaction during everyday activities. The MAETS includes 8 components: participation and a productive role; predictable activities; language that follows the child's focus of attention; child initiations; balance of communicative turns; messages to support child comprehension; verbal and nonverbal models; and appropriate expectations and demands. Each component is scored on a 4-point scale where 0 = Absent, 1 = Emerging, 2 = Practicing, and 3 = Mastery. Total scores range from 0 to 32 and higher scores indicate that the level of parent support is better.
Social Communication Change | Baseline and 6, 12, and 18 months thereafter
  The Brief Observation of Social Communication Change (BOSCC) is designed to measures change during treatment in social communication behaviors in young children with ASD. The BOSCC will be coded from a standardized 10-minute video observations of free-play interactions between the child and caregiver collected during clinical assessments.
Intervention Strategy Use | Baseline and 6, 12, and 18 months thereafter
  The Measure of NDBI Strategy Implementation-Caregiver Change (MONSI-CC) measures changes in caregivers' use of core NDBI strategies during parent-mediated early interventions. The MONSI-CC will be independently coded from the same standardized 10-minute parent-child interaction collected as part of the BOSCC and will be examined as a possible mediator of change in BOSCC outcomes.
Observation of Diagnostic Features of Autism Change | Baseline and 3, 6, 9, 12, 15, and 18 months thereafter
  Features of autism spectrum disorder (ASD) will be periodically measured using the Systematic Observation of Red Flags (SORF) of ASD. The SORF is measured from a home observation of everyday activities. The SORF includes 11 red flags in social communication and social interaction and 11 red flags in restricted and repetitive behaviors using the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) diagnostic features rated on a 3 point scale. The total number of red flags ranges from 0 to 22 and higher scores indicate more red flags of ASD. The total composite score ranges from 0 to 66 and higher scores indicate more diagnostic features of ASD.

SECONDARY OUTCOMES:
Autism Symptoms | Baseline and 6, 12, and 18 months thereafter
  Autism symptoms will be measured with the Autism Diagnostic Observation Schedule (ADOS), Second Edition, the gold standard diagnostic measure of ASD. The revised algorithms forming Social-Affect and Restricted Repetitive Behavior ratings of autism symptoms will be used. Scores range from 1 to 10 and higher scores indicate more autism symptoms. A total of score of 1 to 3 indicates no signs of ASD, a score of 4 or 5 suggests that the child may have ASD, while a score of 6 to 10 is indicative of ASD.
Developmental Level | Baseline and 6, 12, and 18 months thereafter
  This study will use four scales of the Mullen Scales of Early Learning (MSEL) to measure developmental level: Fine Motor; Visual Reception; Expressive Language; and Receptive Language. The average of the four cognitive scales forms an Early Learning Composite. The 4 cognitive scales are measured with T scores that range from 10 to 90 based on a mean T score of 50. A higher T score indicates a better developmental level for the child's age. The Early Learning Composite is measured with Standard scores that range from 40 to 160 based on a mean standard score of 100. A higher standard score indicates a better developmental level for the child's age.
Adaptive Behavior | Baseline and 6, 12, and 18 months thereafter
  Adaptive Behavior will be measured with the Vineland Adaptive Behavior Scales, 3rd edition (VABS-3). The VABS-3 provides a standard score in four domains: Communication, Daily Living Skills, Socialization, and Motor Skills. The domain scores are averaged to form an Adaptive Behavior Composite score. The domain and composite standard scores range from 40 to 160 based on a mean standard score of 100. A higher domain and composite standard score indicates a better adaptive behavior for the child's age.
Brief Observation of Autism Symptoms | Baseline and 6, 12, and 18 months thereafter
  The Autism Diagnostic Observation Schedule (ADOS-2) provides a way for clinicians to observe the social communicative behavior and play/imagination of a participant in a relatively natural context and to place these observations within a framework of standardized codes. However, the ADOS-2 is not appropriate to administer via telehealth nor when the parties involved are wearing face masks. Thus, the Brief Observation of Symptoms of Autism (BOSA) provides a context of activities that can be presented by an examiner (e.g., a caregiver, therapist) within a 12-14-minute observation to help fill the gap left by not being able to carry out a valid ADOS. Clinicians familiar with the ADOS-2 can observe the BOSA live, through telehealth, or on recorded video and complete many of the ADOS-2 codes. The ADOS-2 codes will then be used to denote evidence of symptoms of autism and recorded within a DSM-5 checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Wetherby, PhD, Principal Investigator — Florida State University
Locations (8):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - Florida State University Autism Institute, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Weill Cornell Medical College, White Plains, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: Baby Navigator — https://www.babynavigator.com
- See also: Autism Navigator — https://www.autismnavigator.com